CLINICAL TRIAL: NCT01937221
Title: Novel Retinal Imaging Biomarkers in Early Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Duke Institute for Brain Sciences (Unknown); Alzheimer's Association (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00047227
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2017-12

CONDITIONS: Mild Cognitive Impairment; Mild to Moderate Cognitive Impairment
Keywords: mild cognitive impairment; mild to moderate cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- mild cognitive impairment
  Interventions: Other: spectral-domain optical coherence tomography (SD-OCT)
- mild to moderate cognitive impairment
  Interventions: Other: spectral-domain optical coherence tomography (SD-OCT)
- normal or control group
  Interventions: Other: spectral-domain optical coherence tomography (SD-OCT)

INTERVENTIONS:
Other: spectral-domain optical coherence tomography (SD-OCT) — Intervention same to all groups.

SUMMARY:
The goal of this study is to create new retinal imaging processing software useful for the development of novel retinal biomarkers of cognitive impairment associated with Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Result of the standard neuropsychological assessment
2. Are men or postmenopausal women, at least 55 years of age. Postmenopausal women are defined as women who have had a hysterectomy and/or bilateral oophorectomy; or who have been amenorrheic for at least 2 years;
3. Fluency in English
4. Participants in mild cognitive impairment (MCI)/prodromal and mild-to-moderate dementia groups must assign a surrogate for purposes of informed consent and help with protocol compliance.

Exclusion Criteria:

1. Known or suspected diagnosis of non-AD, associated dementia;
2. Major ophthalmologic comorbidities: Ruptured globe, retinal vascular occlusive disease, retinal artery occlusion, anterior ischemic optic neuropathy, media opacification due to corneal abnormalities or cataract that prevent ocular and OCT examination, glaucoma, wet (neovascular) age-related macular degeneration, history of intravitreal injections, and macular edema. If two eyes satisfy the inclusion criteria, both eyes will be included in the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal controls and patients with mild, mild to moderate cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Nerve fiber layer/ganglion cell layer (NFL/GCL) abnormality score | Baseline
  The study will determine the significance of difference in NFL/GCL score between the AD subject groups at baseline.
NFL/GCL abnormality score | 12 months
  The study will determine the significance of difference in NFL/GCL score between the AD subject groups at baseline. Dependent on baseline results, some subjects may have the opportunity to have another measurement taken at 12 months.

SECONDARY OUTCOMES:
Drusen/plaque score | Baseline
  The study will determine the significance of difference in peripheral drusen/amyloid plaque score between the AD subject groups at baseline.
Drusen/plaque score | 12 months
  The study will determine the significance of difference in peripheral drusen/amyloid plaque score between the AD subjects groups at baseline. Dependent on baseline results, some subjects may have the opportunity to have a second measurement at 12 months.
Total drusen area | Baseline
  The study will determine the significance of difference in total drusen area between the AD subject groups at baseline.
Total drusen area | 12 months
  The study will determine the significance of difference in total drusen area between the AD subject groups at baseline. Dependent on baseline results, some subjects may have the opportunity to have a second measurement taken at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Whitson, MD, MHS, Principal Investigator — Duke University; Eleonora Lad, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States